CLINICAL TRIAL: NCT03075436
Title: The Impact of Enhanced, Demand-side Sanitation and Hygiene Promotion on Sustained Behavior Change and Health in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Emory Ethiopia (Unknown); Amhara Regional Health Bureau (Unknown); Federal Democratic Republic of Ethiopia Ministry of Health (Unknown)
Responsible Party: Principal Investigator, Matthew Freeman, MPH, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00076141
Record Dates: First submitted 2017-03-07; First posted 2017-03-09 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Sustained Behavior Change; Mental Well-being
Keywords: Sanitation; Hygiene; Public Health; Behavior change; Neglected tropical diseases; Demand-side sanitation and hygiene; Mental well-being; Water insecurity; Sanitation insecurity; Collective efficacy
MeSH Terms: conditions — Psychological Well-Being; Neglected Diseases | interventions — Hygiene; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced demand-side sanitation, hygiene (Experimental): The intervention group will receive a package of enhanced, demand-side sanitation and hygiene interventions that are informed by formative research and facilitated by local government and Emory Ethiopia partners.
  Interventions: Behavioral: Enhanced demand-side sanitation, hygiene
- Standard of care (Active Comparator): The comparison group will receive the current standard of care, including potential implementation of government-led policies and programs.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Enhanced demand-side sanitation, hygiene — The enhanced, demand-side sanitation and hygiene intervention package will be informed by findings from formative research, and will consist of interventions designed to enhance sanitation and hygiene messaging to better facilitate behavior change, and intensify implementation of related community-based interventions via engagement of various delivery modalities.
  Arms: Enhanced demand-side sanitation, hygiene
Behavioral: Standard of care — The comparison group will receive the current standard of care, including potential implementation of government-led policies and programs.
  Arms: Standard of care

SUMMARY:
This study is a two-year evaluation investigating the impacts of an enhanced, demand-side sanitation and hygiene intervention on sustainable adoption of improved water, sanitation, and hygiene (WASH) practices and mental well-being.

DETAILED DESCRIPTION:
This study utilizes a cluster randomized, controlled trial design to examine the impacts of an enhanced, demand-side sanitation and hygiene intervention on behavior change and health in Amhara, Ethiopia. The study will test hypotheses set out in the investigation team's theory of change through the measurement and evaluation of process indicators, intermediate and shorter-term behavioral outcomes, and longer-term behavioral and health impacts, including mental well-being.

The study aims to: (1) identify ways in which WASH-related behavior change components preventive for neglected tropical diseases (NTDs) can be mainstreamed into the government-led Health Extension Program; (2) document the effectiveness of an enhanced demand-side sanitation and hygiene intervention; (3) investigate whether changes in personal hygiene, sanitation, and water behaviors are sustained; (4) document the cost-effectiveness of integrated WASH-related NTD-preventive behavior change promotion; and (5) assess whether collective efficacy and water security modify intervention effectiveness.

ELIGIBILITY:
Inclusion criteria:

* Households residing in kebeles in select woredas of Amhara National Regional State
* Households with at least one adult (18 years of age or older) who provides consent to serve as the survey respondent
* Households with at least one child aged 1-9 years (at baseline) living in the household and consenting to enrollment in the study, including study staff observation of children, specifically their faces and hands

Exclusion criteria:

* Households that refuse to provide consent to enroll in the study or have one adult consent to serve as the survey respondent
* Households that are repeatedly vacant or do not have an appropriate member of the household home to serve as the household's respondent (capable adult 18 years or older) after three attempts within the course of one day (for study enrollment and baseline)
* Households that do not have a household member aged 0-5 years of age (at baseline) living in the household

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10375 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Sustainability of WASH-related behaviours, including NTD-preventive WASH behavior measures | Endline (Up to two years)
  Sustainability of WASH-related behaviors, as measured through changes in the proportion of individuals and households practicing targeted improved NTD-preventive WASH behaviors.
Mental well-being measures | Up to two years
  Mental well-being, as measured through the changes in mental well-being scale scores

SECONDARY OUTCOMES:
Shorter-term behavioral outcome measures | Up to two years
  Proportion of households with improved or shared, but otherwise improved household latrine and washing facilities that are functional and available for use; proportion of households using functional latrines and washing facilities; proportion of households with all members exclusively using a latrine for defecation purposes; proportion of households disposing of child feces in an improved latrine; proportion of households with all children in the household with a clean face and hands.
Intermediate behaviour change antecedent measures | Up to two years
  Proportion of households with improved knowledge regarding the implications of improved WASH practices; proportion of households that indicate positive attitudes, perceptions toward improved sanitation and good hygiene practices; change in normative beliefs and behaviors related to open defecation, exclusive latrine use for defecation, and personal hygiene practices.
Water insecurity measures | Up to two years
  Water insecurity, as measured through changes in water insecurity scale scores
Sanitation insecurity measures | Up to two years
  Sanitation insecurity, as measured through changes in sanitation insecurity scale scores
Collective efficacy measures | Up to two years
  Collective efficacy, as measured through changes in collective efficacy scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Freeman, PhD, Principal Investigator — Emory University
Locations (1):
- Amhara, Amhara National Regional State, Ethiopia

REFERENCES:
- [Derived] Freeman MC, Delea MG, Snyder JS, Garn JV, Belew M, Caruso BA, Clasen TF, Sclar GD, Tesfaye Y, Woreta M, Zewudie K, Gobezayehu AG. The impact of a demand-side sanitation and hygiene promotion intervention on sustained behavior change and health in Amhara, Ethiopia: A cluster-randomized trial. PLOS Glob Public Health. 2022 Jan 7;2(1):e0000056. doi: 10.1371/journal.pgph.0000056. eCollection 2022. PMID 36962125
- [Derived] Delea MG, Snyder JS, Belew M, Caruso BA, Garn JV, Sclar GD, Woreta M, Zewudie K, Gebremariam A, Freeman MC. Design of a parallel cluster-randomized trial assessing the impact of a demand-side sanitation and hygiene intervention on sustained behavior change and mental well-being in rural and peri-urban Amhara, Ethiopia: Andilaye study protocol. BMC Public Health. 2019 Jun 21;19(1):801. doi: 10.1186/s12889-019-7040-6. PMID 31226957